CLINICAL TRIAL: NCT00279071
Title: Use of Acupuncture for Stimulation of Labour
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: exhausted personel after a long recruiting period
Sponsor: Herning Hospital (Other)
Collaborators: Ringkjøbing County Research Fond (Unknown); Union of Midwives Research Fond (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-Modlock; NCT00279071
Record Dates: First submitted 2006-01-18; First posted 2006-01-19 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-07

CONDITIONS: Dystocia
Keywords: dystocia; stimulation; acupuncture; oxytocin
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Acupuncture og acupressure when diagnosed with dystocia — Acupuncture points: sp6 li4 ki3 ki6 bl60 Acupressure points: bl67

SUMMARY:
Hypothesis:Acupuncture can be used as stimulation of labour in case of primary og secondary inertia.

A randomized controlled trial including 150 pregnant women Acupuncture has become a natural part of the range of obstetric treatments offered in danish delivery wards, but there is only little evidence to the effect of the acupuncture.

The women are randomized into to groups.

1. Acupuncture, Acu.points: KI3, Ki6, SP6, BL60, LI4, BL67(acupressure)
2. No treatment

The women will be asked in case beginning signs of inertia, if they want to parcipitate in the trial.

Inclusion criteria:

1. Normal pregnancy
2. In labour (orificium < 8 cm), 37th week or thereafter
3. Ruptured membranes
4. Primary or secondary inertia

The women will just before randomization be vaginally explored and fetal heart monitored. The meassure of effect happens two hours after randomization.

The midwife who measures the effect, is blinded to the treatment or lack of, and also on the including exploration.

Secondary effect meassures: length of labour, use of oxytocin and number of contracions pr/min meassured twice:

1. before the randomization and again 1 hour after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Normal pregnancy
2. In labour (orificium < 8 cm), 37th week or thereafter
3. Ruptured membranes
4. Primary or secondary inertia -

Exclusion Criteria:

1. Pathological pregnancy
2. Pathological labour
3. Medical diseases
4. Women who do not speak and undrestand danish

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-10; Study Completion 2007-03 (Actual)

SECONDARY OUTCOMES:
use of oxytocin | additional need for oxytocin infusion in 1. stage and 2. stage
number of contractions/30 minutes | number og contractions in 1st. stage and 2nd. stage

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Rasmussen, obst. dr.med, Study Chair — Obstetric ward Herning and Holstebro hospitals